CLINICAL TRIAL: NCT01106872
Title: A Pilot Study Targeting Angiogenesis Using Bevacizumab Combined With Chemotherapy and Histone Deacetylase Inhibitor (Valproic Acid) in Advanced Sarcomas
Brief Title: Bevacizumab, Chemotherapy and Valproic Acid in Advanced Sarcomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mohammed M Milhem (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Mohammed M Milhem, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200911736; AVF4761s (Other: UIowa IRB 01)
Record Dates: First submitted 2010-03-22; First posted 2010-04-20 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Sarcoma; Soft Tissue Sarcoma; Locally Advanced Sarcoma; Unresectable Sarcoma; Metastatic Sarcoma
Keywords: Sarcoma; Soft Tissue Sarcoma; Locally Advanced Sarcoma; Unresectable Sarcoma; Metastatic Sarcoma; Valproic Acid; Bevacizumab; Histone Deacetylase Inhibitor
MeSH Terms: conditions — Sarcoma | interventions — Bevacizumab; Gemcitabine; Docetaxel; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Bevacizumab Combined with Gemcitabine, Docetaxel and Valproic Acid in Advanced Sarcoma
  Interventions: Drug: Bevacizumab, Gemcitabine, Docetaxel and Valproic Acid

INTERVENTIONS:
Drug: Bevacizumab, Gemcitabine, Docetaxel and Valproic Acid
  Other Names: Avastin; Gemzar; Taxotere; Depakene; Stavzor

SUMMARY:
The purpose of this study is to test the combination of the chemotherapy drugs Gemcitabine, bevacizumab, and docetaxel with valproic acid to treat patients with metastatic sarcoma. Valproic acid is used by people who have seizures to prevent seizures from happening; however, its use in cancer is investigational. This study will help define the proper dosing of this valproic acid. We will assess the safety of valproic acid with the combination of the above chemotherapy drugs and check for possible side effects. Valproic acid may improve the function of the chemotherapy drugs against the cancer.

DETAILED DESCRIPTION:
Soft tissue sarcomas (STS) are a heterogeneous group of benign and malignant tumors of various supportive tissues arising from the mesoderm. There are 56 known subtypes classified by the tissue of origin. Soft tissue sarcomas account for 1% of all human malignancies. These tumors share a common mesenchymal origin with the vasculature. Many of the signaling pathways involved in angiogenesis also drive sarcoma tumor cell growth. Autocrine and paracrine vascular endothelial growth factor (VEGF) - and platelet-derived growth factor (PDGF)-mediated growth plays a role in the pathogenesis of several sarcoma subtypes1. Despite promising preclinical data supporting a role for angiogenesis inhibition in sarcoma, relatively few clinical trials have evaluated antiangiogenic therapy in sarcoma.

Most of the studies for the use of anti-angiogenic drugs have been taken from phase I trials of refractory solid tumors showing a lack of response in sarcomas. This may be due to an inadequate dose, wrong sequence of the treatment or lack of studies with combination treatments. Given the heterogeneity of sarcomas there may be a benefit in certain subgroups that can easily be missed. A recent clinical trial has shown improved cytotoxic cell kill and response rates by epigenetically modifying the tumor environment prior to chemotherapy. It is believed that the efficacy of angiogenesis inhibitors has been shown to be greatly improved when they are combined with other anticancer drugs.

Tumor metastasis is highly dependent on angiogenesis progressing through a metastatic cascade that includes primary tumor growth, modification of tumor cell growth and behavior and formation of new blood vessels. This angiogenic switch is believed to be the result of changes in the balance of angiogenesis stimulators, inhibitors and modulators present at the site of the tumor growth. These changes are due to both genetic alterations involving RAS, RAF, MYC, SRC, EGFR and HER-2 and tumor suppressor genes and epigenetic circumstances such as hypoxia, inflammation or hormonal stimulation. It is clear that vascular endothelial growth factor (VEGF) has emerged as the key stimulatory molecule for promoting angiogenesis in a variety of human malignancies. Other pro-angiogenic factors can be induced or amplified in the presence of hypoxia hypoglycemia, inflammatory cytokines and altered cell-cell contact. Thus it would be of interest to combine epigenetic modifiers like Valproic acid, a histone deacetylase inhibitor, with Bevacizumab, an anti-angiogenic agent against VEGF and standard chemotherapy (Gemcitabine /docetaxel) to better modulate the cytotoxic effects against sarcomas.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 18 years old.
2. ECOG Performance Status of ≤ 2.
3. Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed.
4. Patients must meet the following laboratory criteria:

   Hematology: Neutrophil count of > 1500/mm3; Platelet count of >100,000/mm3L; Hemoglobin ≥ 9 g/dL Biochemistry:AST/SGOT and ALT/SGPT ≤ 2.5 x upper limit of normal (ULN) or ≤ 5.0 x ULN if the transaminase elevation is due to disease involvement; Serum bilirubin ≤ 1.5 x ULN; Serum creatinine ≤ 1.5 x ULN or 24-hour creatinine clearance ≥ 50 ml/min; Total serum calcium (corrected for serum albumin) or ionized calcium ≥ LLN; Serum potassium ≥ LLN; Serum sodium ≥ LLN; Serum albumin ≥ LLN or 3g/dl; Patients with any elevated alkaline phosphatase due to bone metastasis can be enrolled
5. Screening EKG with a QTc less than 450 msec confirmed by central laboratory prior to enrollment to the study.
6. Baseline MUGA or ECHO done only in subjects with prior doxorubicin exposure. The test must demonstrate LVEF ≥ the lower limit of the institutional normal.
7. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first administration of study treatment and must be willing to use two methods of contraception one of them being a barrier method during the study and for 3 months after last study drug administration
8. Any patient with the diagnosis of locally advanced, unresectable or metastatic sarcoma from any site. These include untreated patients or those treated with chemotherapy 1st line, 2nd line and 3rd line. Patients must have measurable disease defined as at least 1 lesion ≥ 1cm in the greatest dimension.
9. Previous exposure to Gemcitabine and Taxotere will only be allowed if there is no residual toxicity from previous treatments. Toxicity must be graded as 0 or 1 prior to study.
10. Patients must have had disease progression on or following their most recent treatment regimen or on presentation for the first time with locally advanced unresectable or metastatic disease.

1.All subtypes of sarcoma are eligible for the trial.

Exclusion Criteria:

1. Prior use of Bevacizumab for the treatment of cancer.
2. Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer.
3. Patients who will need valproic acid for any medical condition .
4. Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure > 100 mmHg).
5. Prior history of hypertensive crisis or hypertensive encephalopathy.
6. New York Heart Association (NYHA) Grade II or greater congestive heart failure.
7. History of myocardial infarction or unstable angina within 6 months prior to Day 1.
8. History of stroke or transient ischemic attack within 6 months prior to Day 1.
9. Known CNS disease, except for treated brain metastasis: Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, LINAC, or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded.
10. Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
11. History of hemoptysis (>/= 1/2 teaspoon of bright red blood per episode) wit hin 1 month prior to Day 1
12. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
13. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
14. History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
15. Serious, non-healing wound, active ulcer, or untreated bone fracture
16. Proteinuria as demonstrated by a UPC ratio >/= 1.0 at screening
17. Pregnancy (positive pregnancy test) or lactation. Use of effective means of contraception (men and women) in subjects of child-bearing potential
18. Concomitant use of drugs with a risk of causing torsades de pointes
19. Concomitant use of CYP3A4 inhibitors
20. Other concurrent severe and/or uncontrolled medical conditions
21. Patients who have received chemotherapy or any investigational drug < 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
22. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study.
23. Concomitant use of any anti-cancer therapy or radiation therapy.
24. Male patients whose sexual partners are WOCBP not using a double method of contraception during the study and 3 months after the end of treatment. One of these methods must be a condom.
25. Patients with a history of another primary malignancy within 2 years other than curatively treated CIS of the cervix, or basal or squamous cell carcinoma of the skin
26. Patients with known positivity for human immunodeficiency virus (HIV); baseline testing for HIV is not required
27. Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent
28. Bone sarcoma is excluded
29. Patients who are on drugs that prolong QT-interval on EKG (many antiarrhythmics, tricyclics, phenothiazines, and others)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-08-22 (Actual)

PRIMARY OUTCOMES:
Evaluate toxicities | After one cycle (3 weeks)
  Dose-limiting toxicities per CTCAE 4.0; grade 4 hematologic toxicity; grade 3 or 4 hepatotoxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Milhem, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No